CLINICAL TRIAL: NCT01913418
Title: Clinical Efficacy and Serum Proteomic Profiling of Traditional Chinese Medicine, Suan-Zao-Ren Tang, for Sleep Disturbance During Methadone Maintenance: Study Protocol for a Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Clinical Efficacy and Serum Proteomic Profiling of Suan-Zao-Ren Tang for Sleep Disturbance During Methadone Maintenance
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: China Medical University, Taiwan (Other)
Responsible Party: Principal Investigator, Yuan-Yu Chan, Graduate Institute of Integrated Medicine,China Medical University, China Medical University, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NSC 102-2320-B-039-024-
Record Dates: First submitted 2013-07-28; First posted 2013-08-01 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2014-03

CONDITIONS: Opiate Dependence
Keywords: Traditional Chinese Medicine; Suan-Zao-Ren Tang; Methadone; Opiate dependence; Sleep
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Suan-Zao-Ren Tang (Active Comparator): The SZRT formula used in this study is manufactured as a herbal extract powder from the good manufacturing procedures (GMP) of the certified company Kaiser Pharmaceutical Co., Ltd. (Taiwan). Granules were packed in aluminum foil packages and administered orally at a dose of 4 g, three times per day for four weeks.
  Interventions: Drug: Suan-Zao-Ren Tang
- Suan-Zao-Ren Tang placebo (Placebo Comparator): The Suan-Zao-Ren Tang placebo granules are prepared with 4 g starch inside the same colored and sized foil packages.
  Interventions: Drug: Suan-Zao-Ren Tang placebo

INTERVENTIONS:
Drug: Suan-Zao-Ren Tang — SZRT is composed of five herb ingredients as follows: Semen Zizyphi Spinosae (Suanzaoren), Sclerotium Poriae Cocos (Fuling), Radix Ligustici Chuanxiong (Chuanxiong), Rhizoma Anemarrhena (Zhimu), and Radix Glycyrrhizae (Gancao).The SZRT granules were packed in aluminum foil packages and administered orally at a dose of 4 g, three times per day for four weeks.
  Arms: Suan-Zao-Ren Tang
Drug: Suan-Zao-Ren Tang placebo — The Suan-Zao-Ren Tang placebo granules are prepared with 4 g starch inside the same colored and sized foil packages.
  Arms: Suan-Zao-Ren Tang placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of Suan-Zao-Ren Tang in improving sleep quality, anxiety, depression, and heroin craving among methadone-maintained persons with sleep complaints.

DETAILED DESCRIPTION:
Background:

Heroin dependence is one of the major health issues worldwide. Methadone Maintenance Therapy (MMT) is an effective treatment for opioid dependence, but more than three quarters of persons receiving MMT report sleep complaints. Traditional Chinese Medicine (TCM) is one of the most common complementary therapies offered to insomnia patients in Taiwan. Investigators designed a randomized, double-blind, placebo-controlled clinical trial to evaluate the efficacy of TCM in methadone-maintained persons with sleep disturbance.

Methods/design:

In this study, inclusion criteria are persons receiving MMT for at least one month, more than 20 years old, complain insomnia with a Pittsburgh Sleep Quality Index (PSQI) of six or higher. Exclusion criteria include being pregnancy, had serious physical or mental illness, current use (last 30 days) of TCM, had received any antidepressant or neuroleptic medication and inability to read and fill out the forms for the study. The patients were separated into an intervention group (Suan-Zao-Ren Tang, SZRT) and a placebo group for four weeks using a randomized, double-blind procedure. Outcome measures will be assessed at baseline, 4 weeks and 8 weeks after receiving medication. PSQI was used to assess sleep quality over the past 30 days, anxiety and depression levels measured by the Beck Anxiety Inventory (BAI) and Beck Depression Inventory II (BDI-II) were also conducted, heroin craving degree was evaluated by the change of the visual analog scale (VAS). Serum proteins will be detected using a proteomics method based on two-dimensional gel electrophoresis, and the specificity of proteins will confirmed by western blotting. T-test and chi-square tests are used for statistical analysis.

Discussion:

SZRT is a combination of Semen Zizyphi Spinosae (Suanzaoren), Sclerotium Poriae Cocos (Fuling), Radix Ligustici Chuanxiong (Chuanxiong), Rhizoma Anemarrhena (Zhimu), and Radix Glycyrrhizae (Gancao). It was the most commonly prescribed Chinese herbal formula used for the treatment of insomnia. In the classical literature and previous studies, SZRT was said to calm the nerves and nourish the blood to eventually bring on a tranquillizing sensation and improved the quality of sleep without generating significant side effects. In order to evaluate the efficacy of SZRT for sleep disturbance during methadone maintenance, investigators designed a randomized, double-blind, placebo-controlled trial and perform the proteomic-system biology analysis to find the biomarker associated with sleep condition.

ELIGIBILITY:
Inclusion Criteria:

* aged over 20 years
* patients fulfilled the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition criteria for opiate dependence
* patients had been receiving MMT for more than one month
* patients have sleep disturbance complains and with Pittsburgh sleep quality index (PSQI) of greater than six
* Must be able to signed informed consent

Exclusion Criteria:

* had received any antidepressant or neuroleptic medication
* had received any TCM treatment during the previous 30 days
* had any serious physical or mental illness
* had a significant risk of suicide
* pregnancy
* inability to read and fill out the forms for the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2013-07; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
sleep quality | The patients will complete the questionnaire at baseline (first visit), four weeks later (second visit), and eight weeks later (third visit).
  The primary outcome measure under study is the sleep quality. Sleep quality will be assessed using the Taiwanese version of the PSQI, which has demonstrated reliability and validity. It evaluates sleep disturbances in 7subscales: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication and daytime dysfunction. Each subscale is rated on a 4-point scale (0 to 3, with 3 indicating a more profound effect), which is summed together to yield a global score (0to21).

SECONDARY OUTCOMES:
severity of heroin craving | The patients will complete the questionnaire at baseline (first visit), four weeks later (second visit), and eight weeks later (third visit).
  The severity of heroin craving was assessed using a 100 millimeters visual analog scale (VAS).
Beck Anxiety inventory (BAI) | The patients will complete the questionnaire at baseline (first visit), four weeks later (second visit), and eight weeks later (third visit).
  This measure lists 21 symptoms of anxiety such as feeling hot, scared or nervous. Participants will be instructed to rate how much each of these symptoms bothered them in the past week. Each item can be rated on a 4 point Likert scale, ranging from 0 (Not at all) to 3 (Severely) yielding a maximum total score of 63 points.
Beck Depression Inventory (BDI-II, second edition) | The patients will complete the questionnaire at baseline (first visit), four weeks later (second visit), and eight weeks later (third visit).
  Depression symptoms will be measured with the BDI-II. This measure consists of 13 items to evaluate depression, and each item is rated from 0 to 3 according to the degree by which it reflects a patient's state during the previous week. The BDI has a high reliability, and concurrent validity.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of psychiatry, Armed Forces Tao-Yuan General Hospital, No.168 Zhong-Xing Road, Taoyuan, Taiwan, Taoyuan District, Taiwan